CLINICAL TRIAL: NCT03041012
Title: Early Administration of Latency Reversing Therapy and Broadly Neutralizing Antibodies to Limit the Establishment of the HIV-1 Reservoir During Initiation of Antiretroviral Treatment - a Randomized Controlled Trial
Brief Title: Early Administration of Romidepsin and 3BNC117 in Treatment-naïve HIV Patients Starting ART
Acronym: eCLEAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Herning Hospital (Other); Hammersmith Hospitals NHS Trust (Other); St Mary's Hospital, London (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: eCLEAR-001; 2015-002234-53 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-02-02 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hiv
Keywords: HIV-1; Latency Reversal Agent; Immunotherapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — romidepsin; 3BNC117 antibody; Broadly Neutralizing Antibodies; Anti-Retroviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- antiretrovirals (Placebo Comparator): Standard of care
  Interventions: Drug: Antiretrovirals
- antiretrovirals + romidepsin (Active Comparator): Standard of care + LRA
  Interventions: Drug: Romidepsin; Drug: Antiretrovirals
- antiretrovirals + 3BNC117 (Active Comparator): Standard of care + bNAb
  Interventions: Drug: 3BNC117; Drug: Antiretrovirals
- antiretrovirals + romidepsin + 3BNC117 (Active Comparator): Standard of care + LRA + bNAb
  Interventions: Drug: Romidepsin; Drug: 3BNC117; Drug: Antiretrovirals

INTERVENTIONS:
Drug: Romidepsin — 5mg/m2 romidepsin will be administered IV on days 10, 17, and 24 after initiating ART
  Other Names: Istodax
  Arms: antiretrovirals + romidepsin; antiretrovirals + romidepsin + 3BNC117
Drug: 3BNC117 — 30 mg/kg 3BNC117 will be administered IV on day 7 and 21 after initiating ART
  Other Names: Broadly neutralizing antibody
  Arms: antiretrovirals + 3BNC117; antiretrovirals + romidepsin + 3BNC117
Drug: Antiretrovirals — Combination antiretroviral therapy
  Other Names: ART

SUMMARY:
To evaluate the effect of early viral reactivation by latency reversing agents (LRA) and/or administration of potent broadly neutralizing antibodies (bNAb) on the size of the latent HIV-1 reservoir in treatment naïve HIV-1 patients initiating antiretroviral therapy (ART)

DETAILED DESCRIPTION:
The study will be conducted among ART naïve HIV-1-infected patients.

Subjects will continue ART while receiving LRA romidepsin and/or bNAb 3BNC117.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* CD4+ T cell count >200/µL on last visit prior to study entry
* ART naïve
* Able to give informed consent

Exclusion Criteria:

* Any significant acute medical illness (not including primary HIV infection) in the past 8 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate compliance with study therapy
* The following laboratory values at screening, but the values can be repeated within the screening period, but test results must be available before baseline (day 0) and checked for eligibility:

  * Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  * Serum total bilirubin ≥3 ULN
  * Estimated glomerular filtration rate (eGFR) ≤60 mL/min (based on serum creatinine or other appropriate validated markers)
  * Platelet count ≤100 x10^9/L
  * Absolute neutrophil count ≤1x10^9/L
  * Serum potassium, magnesium, phosphorus outside ≥1.5 ULN/LLN
  * Total calcium (corrected for serum albumin) or ionized calcium ≥1.5 ULN/LLN
  * Hepatitis B or C infection as indicated by the presence of hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
* ECG at screening that shows QTc >450 ms when calculated using the Fridericia formula from either lead V3 or V4 [86]
* Use of:

  * Warfarin or warfarin-derivatives
  * HDACi
  * An agent definitely or possibly associated with effects on QT intervals within 2 weeks of screening
  * Drugs that induce or inhibit CYP3A4 or P-gp
* History of:

  * Clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for Torsades de pointes (e.g. heart failure)
  * Malignancy or transplantation, including skin cancers or Kaposi sarcoma
  * Diabetes mellitus
* Receipt of strong immunosuppressive or systemic chemotherapeutic agents within 28 days prior to study entry
* Known resistance to >2 classes of ART
* Known hypersensitivity to the components of romidepsin, 3BNC117 or their analogues
* Women who are pregnant or breastfeeding, or with a positive pregnancy test during screening or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of non-estrogen containing contraceptions (according to the Danish Medicines Agency guidelines) to avoid pregnancy for the 3 week study period and 4 weeks after study treatment or until undetectable plasma HIV-1 RNA using standard assays
* Males or females who are unwilling or unable to use barrier contraception during sexual intercourse for the 3-week study period, and 4 weeks after study treatment or until undetectable plasma HIV-1 RNA using standard assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Plasma HIV RNA kinetics | 3 months
  Time to undetectable (<20 c/mL)
Quantification of the size of the proviral HIV reservoir | 1 year
  Copies of total HIV-1 DNA per 10⁶ CD4+ T cells as measured by digital droplet PCR
Time to viral rebound during ATI | 12 weeks
  Days from stopping ART to plasma HIV RNA >5,000 on two consecutive measurements

SECONDARY OUTCOMES:
Incidence of treatment emerging events (Safety and tolerability) | 1 year
  Frequence and severity of adverse events (AE), adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR) and suspected unexpected serious adverse reactions (SUSAR).
Quantification of the intact proviral DNA | 1 year
  Intact HIV-1 DNA in CD4+ T cells (copies per million cells) as measured by dd-PCR.
Quantification of HIV mRNA and/or p24 positive cells | 30 days from study entry
  Frequency of mRNA/p24 postive per 1 million CD4+ T cells by FISH-flow
Immune reconstitution | 1 year
  Absolute CD4+ and CD8+ T cell count
Analytic treatment interruption (ATI) study | 64 weeks
  Time to first plasma HIV RNA >5000 c/mL
Impact of pre-ART virus sensitivity to 3BNC117 on ATI outcomes | Baseline and at viral rebound
  3BNC117 sensitivity determined by PhenoSense and/or HIV env sequencing
T cell mediated HIV specific immunity | First of 365 days
  T cell immunity as determined by the HIV AIM assay

OTHER OUTCOMES:
Plasma cytokine and immune activation biomarker levels | 1 year
  Soluble IL-6, sCD14, sCD163

CONTACTS AND LOCATIONS:
Overall Officials: Ole S Søgaard, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (7):
- Denmark (5):
  - Department of Infectious Diseases, Aalborg
  - Dept. of Infectious Diseases, Aarhus University Hospital, Aarhus
  - Department of Infectious Diseases, Copenhagen
  - Department of Infectious Diseases, Hvidovre
  - Department of Infectious Diseases, Odense
- United Kingdom (2):
  - Guy's and St Thomas', London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will be shared following the publication of the primary and secondary endpoints as outlined in this protocol. Data to be shared includes deidentified data points in published, peer-reviewed articles. Additional, related documents will also be available (study protocol, informed consent form). Data will become available following publication with no planned end date.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Individual deidentified participant data (including data dictionaries) will be shared following the publication of the primary and secondary endpoints as outlined in this protocol. Data will become available following publication with no planned end date.
Access Criteria: Access to the data sharing will be given to researchers who provide a methodologically sound proposal for any type of analysis and requires IRB/Ethics committee approval (if applicable). Proposal should be addressed to olesoega@rm.dk.

REFERENCES:
- [Derived] Gunst JD, Pahus MH, Rosas-Umbert M, Lu IN, Benfield T, Nielsen H, Johansen IS, Mohey R, Ostergaard L, Klastrup V, Khan M, Schleimann MH, Olesen R, Stovring H, Denton PW, Kinloch NN, Copertino DC, Ward AR, Alberto WDC, Nielsen SD, Puertas MC, Ramos V, Reeves JD, Petropoulos CJ, Martinez-Picado J, Brumme ZL, Jones RB, Fox J, Tolstrup M, Nussenzweig MC, Caskey M, Fidler S, Sogaard OS. Early intervention with 3BNC117 and romidepsin at antiretroviral treatment initiation in people with HIV-1: a phase 1b/2a, randomized trial. Nat Med. 2022 Nov;28(11):2424-2435. doi: 10.1038/s41591-022-02023-7. Epub 2022 Oct 17. PMID 36253609